CLINICAL TRIAL: NCT03314597
Title: Instrumental or Physical-exercise Rehabilitation of Balance Improve Both Balance and Gait in Parkinson's Disease.
Brief Title: Instrumental or Physical-Exercise Rehabilitation of Balance in Parkinson's Disease? (IPER-PD)
Acronym: IPER-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Antonio Nardone, Professor, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Approval number # 905 CEC
Record Dates: First submitted 2017-10-15; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance exercise group (Active Comparator): Each of the ten sessions was composed of 45 minutes of balance exercises, each treatment being followed by a 15-min final phase of lower limb stretching, performed with the assistance of a physiotherapist. Sessions were repeated two or three times a week, with at least one rest day between one session and the next, over four successive weeks. Each patient was treated on-phase, at the same time of the day across sessions.
  Interventions: Other: Balance exercise
- Mobile platform exercise group (Experimental): Each of the ten sessions was composed of 45 minutes mobile platform training, each treatment being followed by a 15-min final phase of lower limb stretching, performed with the assistance of a physiotherapist. Sessions were repeated two or three times a week, with at least one rest day between one session and the next, over four successive weeks. Each patient was treated on-phase, at the same time of the day across sessions.
  Interventions: Other: Mobile platform exercise

INTERVENTIONS:
Other: Balance exercise — Patients in the balance exercise group received a personalized exercise program developed by an expert physiotherapist. There was no predefined duration for each item of the set of exercises, but all patients underwent an overall 45 min period training per day according to the same schedule. This schedule was based on the Otago Exercise Program and Practice Guidelines for the treatment of Parkinson's disease. Patients did not wear shoes for balance training. All exercises were performed without upper-limb support and with the supervision of a physiotherapist.
  Arms: Balance exercise group
Other: Mobile platform exercise — Patients entered the mobile platform and put on a security harness (no weight unloading), which they wore during the entire session on the platform training. The arms were free to move, but they were asked not to reach out for support. Each patient underwent 45 minutes of training (resting periods included), in which from 6 to 8 perturbation patterns were administered, each one lasting about 4 minutes. During training, the platform moved in the antero-posterior, latero-lateral and diagonal (45 deg) direction with respect to the body. The periodic platform displacement was 10 cm, regardless of the frequency, which could range from 0.3 to 0.6 Hz. Patients stood with eyes open and closed and feet together or 20 cm apart depending on the perturbation subtype.
  Arms: Mobile platform exercise group

SUMMARY:
We hypothesized that rehabilitation specifically addressing balance in Parkinson ́s disease patients might improve not only balance, but locomotion as well. Two balance training protocols (standing on a moving platform, and traditional balance exercises) were compared by assigning patients to two groups: moving platform (n=15) and balance exercises (n=17). Platform moved periodically in antero-posterior, latero-lateral and oblique direction, with and without vision in different trials. Balance exercises were based on Otago Exercise Program. Both platform and exercises sessions were administered from easy to difficult. Outcome measures were: a) balancing behaviour, assessed both by index of stability (IS) on platform and by Mini-BESTest, b) gait, assessed both by baropodometry and by Timed Up and Go (TUG) test. Falls Efficacy Scale-International (FES-I) and Parkinson's Disease Questionnaire (PDQ-8) were administered. Both groups exhibited better balance control, as assessed both by IS and by Mini-BESTest. Gait speed at both baropodometry and TUG also improved in both groups. Scores of FES-I and PDQ-8 showed a marginal improvement. A four-week treatment featuring no gait training, but focussed on challenging balance tasks produces considerable gait enhancement in mildly to moderately affected patients. Walking problems in PD depend on postural instability and are successfully relieved by appropriate balance rehabilitation.

DETAILED DESCRIPTION:
The importance for training balance in connection with rehabilitation aimed at improving gait is easily stressed by considering the complex motor behaviour underpinning more challenging conditions than linear walking, as walking-and-turning, where the turn-related changes in feet, trunk and head movements are integral part of he kinematics of the steering body (Courtine and M. Schieppati, 2003; Crenna et al, 2007). It is no wonder that freezing of gait and increased risk of falling (Schlenstedt et al., 2016) is associated with abnormal bilateral coordination and turning. Hence, the present investigation somehow diverges from the theory of the task-specific training (Bayona et al., 2005), but considers instead the relevance for locomotion enhancement of training balance control, by hypothesising that specific balance rehabilitation might be sufficient for gait improvement. Here, we trained PD patients with two different treatments, both specifically addressing balance. A platform onto which subjects stood moved in antero-posterior, latero-lateral and diagonal direction in the horizontal plane. A simpler moving-platform protocol had been previously exploited for testing and enhancing balance capacities in patients with PD and with vestibular deficit (Nardone et al., 2010; De Nunzio 2007). This platform protocol challenges both the anticipatory and the reactive capacities to the ongoing postural perturbations, thereby training dynamic balance control, aiming at the balance problems encountered during every day activity.

The outcome of the platform treatment was compared to that obtained in another group of matched patients with PD by standardized and validated exercises aimed at training balance and dynamic balance (Renfro et al., 2016). Of note, these exercises contained no dynamic component (i.e. gait-related exercises) of balance training, contrary to Conradsson et al. 2017. Both treatments (platform and exercises) were tailored to the patient individual capacities, and their difficulty gradually increased all along the duration of the treatment (Conradsson et al., 2017). In this context, we estimated any improvement in balance control by indexes of dynamic stability during a balance perturbation test on the mobile platform and by clinical scores related to dynamic balance control. Gait improvement was both evaluated instrumentally and assessed by a functional clinical test.

ELIGIBILITY:
Inclusion Criteria:

* patients with mild to moderate idiopathic Parkinson's disease (PD) (Hoehn-Yahr stage between 1.5 and 3)

Exclusion Criteria:

* orthopaedic conditions restricting exercise, or deep brain stimulation surgery or evidence of dementia . Patients not able walk independently.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2015-12-09 (Actual); Study Completion 2015-12-22 (Actual)

PRIMARY OUTCOMES:
Assessment of balancing behaviour by sinusoidal translation of the supporting platform. | 4 weeks
  The subjects stood upright on a platform that moved continuously 10 cm forward and backward on the horizontal plane at a frequency of sinusoidal translation of 0.4 Hz. The entire test comprised 60 cycles of motion, lasting 2 and a half min. All subjects were blindfolded, their sagittal axis co-planar with the direction of platform movement. Subjects wore a security harness and listened to music through noise-reducing earphones to mask the faint sound produced by the platform mechanism. A physiotherapist stood by the side to support the patient in case of balance loss. Body movements were recorded by detection of 3 reflective markers placed on pterion (head), greater trochanter (hip), and lateral malleolus (invariable with respect to the moving platform). The instantaneous markers' position was recorded by means of a stereometric device (Vicon 460, Oxford Metrics, UK) at a sampling frequency of 120 Hz.
The Mini-Balance Evaluation Systems Test | 4 weeks
  The Mini-Balance 265 Evaluation Systems Test (Mini-BESTest) is a 14-item balance scale that takes 15 min to administer. It specifically addresses dynamic equilibrium, and is highly reliable. Each item is scored on a 3-level ordinal scale from 0 to 2, with 2 representing no impairment and 0 representing severe impairment of balance. The total score ranges from 0 to 28
Assessment of gait performance by baropodometry | 4 weeks
  An electronic walkway (GAITRite®, CIR Systems, Sparta, NJ, USA) returned the baropodometric gait variables. The walkway is 460 cm long, has an area of pressure sensors of 366 cm x 61 cm containing 13824 active sensors, and has a sampling frequency of 80 Hz. The GAITRite system has validity and test-retest reliability in patients with PD. Patients were instructed to walk at their usual velocity. They began walking 2 m before the walkway and continued for 2 m past the end, in order to eliminate acceleration and deceleration events from the acquisition. After one familiarizing trial, the data from four successive trials were recorded. Gait speed, step length and cadence were averaged over the four trials
Timed Up and Go Test (TUG) | 4 weeks
  To evaluate gait in a functional situation of daily living, we used the TUG test. This is a functional measure in which subjects stand up from a chair, walk past a horizontal line marked with tape on the floor at 3 m from start, turn around, walk back and sit down at their comfortable pace . TUG duration greater than 16 s indicates an increased risk of falls in patients with PD. The test has demonstrated an excellent test-retest and inter-rater reliability in PD. Three trials were performed, timed with a stopwatch, and the results obtained from the last two trials were averaged

SECONDARY OUTCOMES:
Fear of Falling | 4 weeks
  In order to evaluate fear of falling, all patients filled the Falls Efficacy Scale-International (FES-I). It is a self-report questionnaire developed for use in elderly populations to assess fear of falling. A series of 16 questions assesses the respondent's fear of falling for a range of ADLs. Each question was rated on a four-point scale from 1 ('not at all concerned' about falls) to 4 ('very concerned').
The Parkinson's Disease Questionnaire (PDQ-8) | 4 weeks
  The Parkinson's Disease Questionnaire (PDQ-8) is an 8-item self-report questionnaire derived from its parent questionnaire, the PDQ-39. It exhibits appropriate levels of reliability, validity and responsiveness. Each item was rated using a five-point scale, corresponding to the frequency with which symptoms occur (from 'never ́ to 'always ́). Total score ranges from 0 to 32. A higher total score reflects a lower health-related quality of life. All patients filled both subjective questionnaires with the aid of a physiotherapist blinded regarding the allocation of the patients.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayona NA, Bitensky J, Salter K, Teasell R. The role of task-specific training in rehabilitation therapies. Top Stroke Rehabil. 2005 Summer;12(3):58-65. doi: 10.1310/BQM5-6YGB-MVJ5-WVCR. PMID 16110428
- [Background] Conradsson D, Nero H, Lofgren N, Hagstromer M, Franzen E. Monitoring training activity during gait-related balance exercise in individuals with Parkinson's disease: a proof-of-concept-study. BMC Neurol. 2017 Jan 31;17(1):19. doi: 10.1186/s12883-017-0804-7. PMID 28143463
- [Background] Courtine G, Schieppati M. Human walking along a curved path. I. Body trajectory, segment orientation and the effect of vision. Eur J Neurosci. 2003 Jul;18(1):177-90. doi: 10.1046/j.1460-9568.2003.02736.x. PMID 12859351
- [Background] Crenna P, Carpinella I, Rabuffetti M, Calabrese E, Mazzoleni P, Nemni R, Ferrarin M. The association between impaired turning and normal straight walking in Parkinson's disease. Gait Posture. 2007 Jul;26(2):172-8. doi: 10.1016/j.gaitpost.2007.04.010. Epub 2007 May 29. PMID 17532636
- [Background] De Nunzio AM, Nardone A, Schieppati M. The control of equilibrium in Parkinson's disease patients: delayed adaptation of balancing strategy to shifts in sensory set during a dynamic task. Brain Res Bull. 2007 Sep 28;74(4):258-70. doi: 10.1016/j.brainresbull.2007.06.020. Epub 2007 Jul 23. PMID 17720548
- [Background] Nardone A, Godi M, Artuso A, Schieppati M. Balance rehabilitation by moving platform and exercises in patients with neuropathy or vestibular deficit. Arch Phys Med Rehabil. 2010 Dec;91(12):1869-77. doi: 10.1016/j.apmr.2010.09.011. PMID 21112428
- [Background] Renfro M, Bainbridge DB, Smith ML. Validation of Evidence-Based Fall Prevention Programs for Adults with Intellectual and/or Developmental Disorders: A Modified Otago Exercise Program. Front Public Health. 2016 Dec 6;4:261. doi: 10.3389/fpubh.2016.00261. eCollection 2016. PMID 27999771
- [Background] Schlenstedt C, Muthuraman M, Witt K, Weisser B, Fasano A, Deuschl G. Postural control and freezing of gait in Parkinson's disease. Parkinsonism Relat Disord. 2016 Mar;24:107-12. doi: 10.1016/j.parkreldis.2015.12.011. Epub 2015 Dec 18. PMID 26762797
- [Derived] Giardini M, Nardone A, Godi M, Guglielmetti S, Arcolin I, Pisano F, Schieppati M. Instrumental or Physical-Exercise Rehabilitation of Balance Improves Both Balance and Gait in Parkinson's Disease. Neural Plast. 2018 Mar 7;2018:5614242. doi: 10.1155/2018/5614242. eCollection 2018. PMID 29706993